CLINICAL TRIAL: NCT03668002
Title: Randomized Trial of Fistula Versus Graft in Elderly Patients Pilot Study (RIGEL Pilot)
Brief Title: Trial of Fistula Versus Graft in Elderly Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to slow recruitment.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Theodore Yuo, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO17100473
Record Dates: First submitted 2018-09-04; First posted 2018-09-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: End Stage Renal Disease; Arteriovenous Fistula; Arteriovenous Graft
Keywords: Fistula vs. Graft
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Arteriovenous Shunt, Surgical

STUDY DESIGN:
Intervention Model Description: This study will provide preliminary data and possibly demonstrate feasibility of a large scale randomized controlled trial comparing AVF and AVG in elderly patients (defined as patients over 65 years of age) receiving hemodialysis through a TDC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arteriovenous Fistula (AVF) (Placebo Comparator): If the participant is randomized to the AVF arm of the trial, the surgeon will connect an artery to a vein in the upper extremity, without using artificial material as conduit.
  Interventions: Procedure: Arteriovenous Fistula (AVF)
- Arteriovenous Graft (AVG) (Active Comparator): If the participant is randomized to the AVG arm of the trial, the surgeon will place a synthetic graft connecting an artery and vein under the skin in an upper extremity.
  Interventions: Procedure: Arteriovenous Graft (AVG)

INTERVENTIONS:
Procedure: Arteriovenous Fistula (AVF) — If the participant is randomized to the AVF arm of the trial, the surgeon will connect an artery to a vein in the upper extremity, without using artificial material as conduit.
  Arms: Arteriovenous Fistula (AVF)
Procedure: Arteriovenous Graft (AVG) — If the participant is randomized to the AVG arm of the trial, the surgeon will place a synthetic graft connecting an artery and vein under the skin in an upper extremity.
  Arms: Arteriovenous Graft (AVG)

SUMMARY:
This open-label pilot randomized controlled trial will test the feasibility and safety of randomizing patients over 65 years old who start hemodialysis with a tunneled dialysis catheter (TDC), and are eligible to receive either arteriovenous fistula (AVF) or arteriovenous graft (AVG), to an AVF strategy (comparator) or to an AVG strategy (intervention). The primary outcome is feasibility, which we will assess by measuring: (1) the proportion of randomized participants who receive the assigned arteriovenous access; and (2) the annual rate of enrollment in the study, accounting for the number of surgeons who participate. Secondary outcomes will include perioperative morbidity and mortality, catheter removal rates, additional procedures performed, and the reasons a patient may not receive the assigned AV access.

DETAILED DESCRIPTION:
End-stage renal disease requiring dialysis affects approximately 400,000 patients in the United States with 100,000 new patients starting dialysis annually. The vast majority of those patients utilize hemodialysis (HD), and of that group, approximately 80% start with a tunneled dialysis catheter (TDC). Current guidelines discourage TDC, due to the risk of serious complications like bloodstream infections, central venous stenosis, and an associated increased mortality risk. The preferred alternative is an arteriovenous (AV) access, either native arteriovenous fistulas (AVF) or prosthetic arteriovenous grafts (AVG). AVF are considered the ideal long-term vascular access due to longer patency, lower costs, and an association with longer survival as compared to AVG when they successfully mature. However, AVF frequently require many months to mature after being constructed and have high primary failure rates (i.e., inability to be used without revision); AVG typically perform better short term, enabling early TDC removal and reduction in catheter related harms, but higher rates of failure and complications long term.

In older populations, multiple studies have suggested that the elderly population may not benefit from AVF as opposed to AVG, due to high AVF primary failure rates and overall abbreviated life expectancy that minimizes any possible long-term benefit with AVF.

METHODS AND ANALYSIS: This open-label pilot randomized controlled trial will test the feasibility and safety of randomizing patients over 65 years old who start hemodialysis with a TDC (the most common initial type of HD access), and are eligible to receive either AVF or AVG, to an AVF strategy (comparator) or to an AVG strategy (intervention). We will enroll 50 patients. Participants will provide informed consent, and they will be assigned to the AVF or AVG arms. The primary outcome is feasibility, which we will assess by measuring: (1) the annual rate of enrollment in the study, accounting for the number of surgeons who participate; and (2) the proportion of randomized participants who receive the assigned AV access. Secondary outcomes will include perioperative morbidity and mortality, catheter removal rates, additional procedures performed, and the reasons a patient may not receive the assigned AV access after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 65 years old.
* On hemodialysis through a tunneled dialysis catheter.
* In the surgeon's opinion, both a fistula and a graft can be reasonably attempted, based on the patient's anatomy.

Exclusion Criteria:

* Unable to provide informed consent.
* Unable to be medically cleared for surgery
* Does not wish to have surgery.
* Does not wish to be randomized.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects that received assigned AV access (AVF vs. AVG) | 12 months
  Adherence to assigned AV access (AVF vs. AVG) during randomization will be measured, expressed as a proportion of all subjects randomized.

SECONDARY OUTCOMES:
Rate of accrual of subjects to the study | 12 months
  Rate of subjects successfully randomized, expressed as subjects per year per surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Yuo, MD MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No